CLINICAL TRIAL: NCT00633906
Title: Reducing HIV Risk in Female Teens: A Tailored Approach
Brief Title: HORIZONS HIV Intervention
Acronym: HORIZONS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ralph J. DiClemente, Principal, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00045957; MH061210 (Other: Other)
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: HIV; Sexually Transmitted diseases; Adolescents; Prevention; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): HORIZONS HIV Intervention. Two-session, group-based interactive intervention.
  Interventions: Behavioral: HORIZONS HIV Intervention
- 2 (Active Comparator): Enhanced standard-of-care session. One hour, video-based and brief discussion.
  Interventions: Behavioral: enhanced standard-of-care

INTERVENTIONS:
Behavioral: HORIZONS HIV Intervention — Two-session, group-based interactive HIV prevention intervention
  Arms: 1
Behavioral: enhanced standard-of-care — 1 hour group session consisting of an HIV prevention video, a question and answer session with an African American woman health educator, and participation in a group discussion about how to avoid acquiring HIV.
  Arms: 2

SUMMARY:
The Horizons Program will test the efficacy of a multi-session HIV prevention program for African American female teens attending reproductive health clinics in Atlanta, GA.

DETAILED DESCRIPTION:
African-American adolescent females are a population at high risk for HIV infection. Recent findings suggest that culturally and gender appropriate HIV interventions can significantly reduce HIV-associated sexual risk behaviors among this vulnerable population. The Horizons HIV intervention was developed for African-American female adolescents attending reproductive health clinics in Atlanta, GA. The specific objectives were:

1. To evaluate the efficacy of the HORIZONS HIV intervention plus standard of care counseling versus the standard of care counseling alone in reducing self-reported HIV sexual risk behaviors and incident STDs over a 12 month follow-up period.
2. To evaluate the cost-effectiveness of the HORIZONS HIV intervention plus standard of care counseling to the standard of care counseling alone with respect to reducing risky sexual behavior and averting incident STDs.

715 participants, ages 15-21, were recruited and enrolled at a large urban county health department, a teen clinic in a public hospital and a reproductive health clinic in the Atlanta area. After a computer interview assessing adolescents' sexual risk and preventive behaviors, and STD testing (Chlamydia and gonorrhea), participants were randomized to one of 2 conditions: the HORIZONS Intervention or the Standard-of-care counseling group. Two trained female health educators lead the 2-session HORIZONS intervention which addressed gender and ethnic pride issues, STD/HIV knowledge, assertive partner communication and refusal skills, and role-play practice. Social Cognitive Theory (SCT) and the Theory of Gender and Power were complementary theoretical frameworks guiding the design and implementation of the HIV intervention. To supplement this group intervention, four phone contacts delivered by the original health educator were conducted during the follow-up period. The supplemental contacts reinforced workshop materials with an individually tailored plan for each participant. The control group received tracking calls only. Follow-up assessments identical to the baseline were conducted at 6 and 12-months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Female
* African American
* Ages 15-21
* Receiving care at participating clinic
* Vaginal sex in the past 60 days
* Ability to give written informed consent

Exclusion Criteria:

* Married
* Pregnant
* In a detention center

Ages: 15 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 715 (Actual)
Dates: Start 2002-04; Primary Completion 2004-08 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Proportion of condom protected vaginal sex acts over the last 60 days | 6 and 12 months post-randomization

SECONDARY OUTCOMES:
Incident infection of chlamydia or gonorrhea as confirmed by laboratory PCR testing | 6 and 12 months post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Ralph J DiClemente, PhD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Fulton County Department of Health and Wellness, Atlanta, Georgia
  - Grady Teen Clinic, Atlanta, Georgia
  - Planned Parenthood of GA, Atlanta, Georgia

REFERENCES:
- [Result] Sales JM, DiClemente RJ, Rose ES, Wingood GM, Klein JD, Woods ER. Relationship of STD-related shame and stigma to female adolescents' condom-protected intercourse. J Adolesc Health. 2007 Jun;40(6):573.e1-6. doi: 10.1016/j.jadohealth.2007.01.007. Epub 2007 Mar 26. PMID 17531767
- [Result] Crosby RA, DiClemente RJ, Wingood GM, Salazar LF, Rose E, Sales JM, Caliendo AM. Oral contraceptive use may not preclude condom use: a study of non-pregnant African-American adolescent females. Sex Transm Infect. 2007 Jun;83(3):216-8. doi: 10.1136/sti.2006.022442. PMID 17569720
- [Result] Woods ER, Klein JD, Wingood GM, Rose ES, Wypij D, Harris SK, Diclemente RJ. Development of a new Adolescent Patient-Provider Interaction Scale (APPIS) for youth at risk for STDs/HIV. J Adolesc Health. 2006 Jun;38(6):753.e1-7. doi: 10.1016/j.jadohealth.2005.08.013. PMID 16730606
- [Result] Spitalnick JS, DiClemente RJ, Wingood GM, Crosby RA, Milhausen RR, Sales JM, McCarty F, Rose E, Younge SN. Brief report: sexual sensation seeking and its relationship to risky sexual behaviour among African-American adolescent females. J Adolesc. 2007 Feb;30(1):165-73. doi: 10.1016/j.adolescence.2006.10.002. Epub 2006 Nov 30. PMID 17140653
- [Result] DiClemente RJ, Wingood GM, Crosby RA, Salazar LF, Rose E, Sales JM, Caliendo AM. Prevalence, correlates, and efficacy of selective avoidance as a sexually transmitted disease prevention strategy among African American adolescent females. Arch Pediatr Adolesc Med. 2008 Jan;162(1):60-5. doi: 10.1001/archpediatrics.2007.5. PMID 18180414
- [Result] Salazar LF, Crosby RA, Diclemente RJ, Wingood GM, Rose E, Sales JM, Caliendo AM. Personal, relational, and peer-level risk factors for laboratory confirmed STD prevalence among low-income African American adolescent females. Sex Transm Dis. 2007 Oct;34(10):761-6. doi: 10.1097/01.olq.0000264496.94135.ac. PMID 17507835
- [Result] Caliendo AM, Jordan JA, Green AM, Ingersoll J, Diclemente RJ, Wingood GM. Real-time PCR improves detection of Trichomonas vaginalis infection compared with culture using self-collected vaginal swabs. Infect Dis Obstet Gynecol. 2005 Sep;13(3):145-50. doi: 10.1080/10647440500068248. PMID 16126499
- [Derived] Rosenbaum JE, Zenilman JM, Rose E, Wingood GM, DiClemente RJ. Semen says: assessing the accuracy of adolescents' self-reported sexual abstinence using a semen Y-chromosome biomarker. Sex Transm Infect. 2017 Mar;93(2):145-147. doi: 10.1136/sextrans-2016-052605. Epub 2016 May 4. PMID 27147615
- [Derived] Swartzendruber A, Brown JL, Sales JM, Murray CC, DiClemente RJ. Sexually transmitted infections, sexual risk behavior, and intimate partner violence among African American adolescent females with a male sex partner recently released from incarceration. J Adolesc Health. 2012 Aug;51(2):156-63. doi: 10.1016/j.jadohealth.2011.11.014. Epub 2012 Feb 28. PMID 22824446
- [Derived] DiClemente RJ, Wingood GM, Rose ES, Sales JM, Lang DL, Caliendo AM, Hardin JW, Crosby RA. Efficacy of sexually transmitted disease/human immunodeficiency virus sexual risk-reduction intervention for african american adolescent females seeking sexual health services: a randomized controlled trial. Arch Pediatr Adolesc Med. 2009 Dec;163(12):1112-21. doi: 10.1001/archpediatrics.2009.205. PMID 19996048